CLINICAL TRIAL: NCT01284348
Title: An Open-Label Randomized, Phase 2A, Dose-Ranging Study of Sotatercept (ACE-011) for Chemotherapy-Induced Anemia in Subjects With Advanced or Metastatic Solid Tumors Treated With Platinum-Based Chemotherapeutic Regimens
Brief Title: To Determine Safe and Effective Dose of Sotatercept for the Treatment of Chemotherapy Induced Anemia in Participants With Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Persistent low enrollment made study continuation no longer feasible
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 7962-015; ACE-011-NSCL-001 (Other: Celgene); 2010-022561-10 (EudraCT Number)
Record Dates: First submitted 2010-12-17; First posted 2011-01-27 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-07

CONDITIONS: Anemia; Carcinoma, Non-Small-Cell Lung; Carcinoma, Small-Cell Lung; Bladder Cancer; Cancer of Head and Neck; Uterine Cervical Cancer
Keywords: Chemotherapy induced anemia; Non-small cell lung cancer
MeSH Terms: conditions — Anemia; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Urinary Bladder Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sotatercept 15 mg (Experimental): Participants will receive sotatercept 15 mg by subcutaneous (SC) injection once every 42 days, up to four doses.
  Interventions: Drug: Sotatercept 15 mg
- Sotatercept 30 mg (Experimental): Participants will receive sotatercept 30 mg by SC injection once every 42 days, up to four doses.
  Interventions: Drug: Sotatercept 30 mg

INTERVENTIONS:
Drug: Sotatercept 15 mg — Sotatercept 15 mg SC injection once every 42 days, up to four doses
  Other Names: ACE-011
  Arms: Sotatercept 15 mg
Drug: Sotatercept 30 mg — Sotatercept 30 mg SC injection once every 42 days, up to four doses
  Other Names: ACE-011
  Arms: Sotatercept 30 mg

SUMMARY:
The purpose of this study was to determine an effective and safe dose of sotatercept (ACE-011) for the treatment of chemotherapy-induced anemia (CIA) in participants with metastatic non-small cell lung cancer (NSCLC) who are being treated with first-line platinum based chemotherapy.

DETAILED DESCRIPTION:
The ACE-011-NSCL-001 Phase 2a study was an open-label, randomized, dose-ranging study designed to assess the efficacy, safety, tolerability, pharmacokinetic and quality of life of sotatercept for treatment of CIA in participants with advanced or metastatic solid tumors treated with platinum-based chemotherapeutic regimens. Other objectives included the effect of sotatercept treatment on bone metabolism, the evaluation of the expression of Activin A and other proteins/biomarkers (including myostatin and follistatin) and the assessment of renal function biomarkers. The study consisted of a Screening Period, a Treatment Period of approximately 6 months (up to 4 doses of sotatercept at either 15 mg or 30 mg administered subcutaneously every 42 days) and a Post-treatment Follow-up Period or End of Treatment (42 days after the last dose of sotatercept). The study was terminated early due to a slower than expected rate of enrollment as a result of substantial changes in the standard of care for cancer participants with anemia which resulted in challenges to timely accrual and completion of the study. Therefore, 26 participants were randomized into the study and the planned Part 2 of the study consisting of a double-blind, randomized, placebo-controlled Phase 2b/3 study conducted at the optimal dose of sotatercept in up to 750 participants with metastatic NSCLC was not performed. Due to the small sample size and variability of the data, changes were made to modify the study endpoints and revise them to be exploratory only.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women >18 years of age
2. Part 1: Histologically confirmed (cytology or biopsy) solid tumor malignancy, excluding those solid tumors treated with curative intent.

   Part 2: Histologically confirmed non-small cell lung cancer
3. Documented metastatic disease
4. Measurable or non-measurable disease evaluable by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
5. All of the following laboratory values:

   * Hemoglobin ≥6.5 to <11.0 g/dL (≥65 to <110 g/L), due to chemotherapy-induced anemia
   * Absolute neutrophil count ≥500/mm^3
   * Platelet count ≥75,000/mm^3 (>2 hours since prior platelet transfusion
   * Adequate renal function

     * creatinine clearance ≥40mL/min or ≥50 mL/min if cisplatin is concomitantly administered and
     * urine protein / creatinine ratio ≤1.0; or ≤2.0 if bevacizumab (Avastin®) is concomitantly administered
   * Hepatic function (bilirubin <1.5 x upper limits of normal (ULN); AST and ALT <3.0 x ULN and ≤5.0 ULN for participants with liver metastases)
6. Participants must have received:

   * at least one cycle and up to 4 cycles (q3w schedule) of platinum-based chemotherapy and be randomized prior to receiving Cycle 5 OR
   * at least one cycle and up to 3 months (depending upon regimen) of platinum-based chemotherapy
7. >28 days since previous treatment with ESA
8. >14 days since last red blood cell transfusions
9. Eastern Oncology Cooperative Group (ECOG) Performance status 0-2
10. For females of childbearing potential, highly effective method of birth control for at least 28 days before starting study, during participation and at least 112 days following last dose of sotatercept
11. Males must use latex condom or non-latex condom not made of (animal) membrane during any sexual contact with female of childbearing potential
12. Life expectancy of >3 months
13. Willing to adhere to study visit schedule
14. Understand and voluntarily sign informed consent

Exclusion Criteria:

Part 2 only, history of prior regimen(s)of platinum-based chemotherapy for metastatic NSCLC and/or history of adjuvant platinum-based chemotherapy with last dose received less than six months prior to the start of current first-line platinum-based chemotherapy for metastatic NSCLC.

1. National Cancer Institute Common Terminology for Adverse Events Grade >3 toxicity
2. Prior radiation to >20% of whole skeleton
3. Prior regimen(s) of platinum based chemotherapy for metastatic disease and/or history of adjuvant platinum-based chemotherapy with the last dose received less than six months prior to the start of current first-line platinum-based chemotherapy for metastatic disease
4. Central nervous system metastases
5. Clinically significant pulmonary, endocrine, neurologic, gastrointestinal, hepatic, or genitourinary disease unrelated to underlying malignancy
6. Classification of 3 or higher heart failure (as classified by New York Heart Association)
7. History of thrombosis, deep vein thrombosis, pulmonary emboli, or embolic stroke, if not stable on anticoagulants and/or one of these events occurring in past 6 months
8. Diagnosis of a myeloid malignancy or known history of myelodysplasia
9. Recent history (within 14 days of Day 1) of IV/oral antibiotics due to post septic episode
10. Uncontrolled hypertension. Controlled hypertension is considered clinically stable, and systolic blood pressure (SBP) must be <150 mmHg and diastolic blood pressure (DBP) must be < 00 mmHg.
11. Known human immunodeficiency virus (HIV)
12. Known active hepatitis B or C antibody
13. Iron deficiency
14. History of anemia as a result of inherited hemoglobinopathy
15. History of anemia due to autoimmune or hereditary hemolysis or gastrointestinal bleeding
16. Received treatment with another investigational drug or device within 28 days prior to Day 1, or if the half life of the previous product is known, within 5 times the half life prior to dosing, whichever may be longer.
17. Any prior use of sotatercept.
18. Pregnant or lactating females or females planning to become pregnant
19. History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product (Refer to the Investigator's Brochure for further information).
20. Major surgery within 30 days prior to Day 1 (participants must have completely recovered from any previous surgery prior to Day 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03-25 (Actual); Primary Completion 2012-09-21 (Actual); Study Completion 2012-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Raftopoulos H, Laadem A, Hesketh PJ, Goldschmidt J, Gabrail N, Osborne C, Ali M, Sherman ML, Wang D, Glaspy JA, Puccio-Pick M, Zou J, Crawford J. Sotatercept (ACE-011) for the treatment of chemotherapy-induced anemia in patients with metastatic breast cancer or advanced or metastatic solid tumors treated with platinum-based chemotherapeutic regimens: results from two phase 2 studies. Support Care Cancer. 2016 Apr;24(4):1517-25. doi: 10.1007/s00520-015-2929-9. Epub 2015 Sep 14. PMID 26370220
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Sotatercept 15 mg: Participants received sotatercept 15 mg by subcutaneous (SC) injection once every 42 days, up to four doses.
- Sotatercept 30 mg: Participants received sotatercept 30 mg by SC injection once every 42 days, up to four doses.
Period: Overall Study
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Started | 14 | 12
Treated | 14 | 11
Completed | 4 | 0
Not Completed | 10 | 12
Not completed — Death | 1 | 1
Not completed — Withdrew consent | 0 | 1
Not completed — Status not recorded | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Sotatercept 15 mg: Participants received sotatercept 15 mg by SC injection once every 42 days, up to four doses.
- Total: Total of all reporting groups
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (14.1) | 68.5 (9.1) | 64.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Hematopoietic Response
Description: A hematopoietic response was defined as an increase in a participant's hemoglobin (Hgb) of ≥1.0 g/dL above the study baseline value for 4 consecutive weeks, in the absence of red blood cell transfusion and/or erythropoiesis-stimulating agents.
Time Frame: Up to Day 28
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 14 | 11
Participants | 2 | 2

2. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to approximately 6 months
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 14 | 11
Participants | 14 | 10

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from date of randomization to date of diagnosis of progressive disease
Time Frame: Up to 6 months
Population: TTP was to be analyzed in Part 2 of the study. Due to low enrollment, the study was terminated early and Part 2 was not performed.
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the start of study drug therapy to the first observation of disease progression or death due to any cause, whichever came first
Time Frame: Up to 12 months
Population: PFS was to be analyzed in Part 2 of the study. Due to low enrollment, the study was terminated early and Part 2 was not performed.
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between randomization and death
Time Frame: Up to 24 months
Population: OS was to be analyzed in Part 2 of the study. Due to low enrollment, the study was terminated early and Part 2 was not performed.
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response was defined as the percentage of participants who achieved an objective confirmed complete (CR) or partial response (PR). Response was determined according to Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 guidelines. CR: The disappearance of all known disease and no new sites or disease-related symptoms confirmed at least 4 weeks after initial documentation. All sites must be assessed, including non-measurable sites, such as effusions, or markers. PR: At least a 30% decrease in the sum of the longest diameters of target lesions, taking as a reference the baseline sum of the longest diameters confirmed at least 4 weeks after initial documentation and no new non-target lesions and/or unequivocal progression of existing non-target lesions. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing.
Time Frame: Up to 12 months
Population: ORR was to be analyzed in Part 2 of the study. Due to low enrollment, the study was terminated early and Part 2 was not performed.
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants Who Experienced an Improvement in Quality of Life Scores
Description: Participants were to be assessed on improvement of quality of life using the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (Version 4.0) and the Lung Cancer Symptom Scale (LCSS). The FACIT Fatigue score ranges from 0 to 52, with 0 representing the best outcome and 52 representing the worst outcome. The LCSS is a 9-item patient-rated scale, 6 of which measure major symptoms (loss of appetite, fatigue, cough, dyspnoea, pain, and haemoptysis), and 3 of which are summation items related to total symptomatic distress, activity, and overall quality of life. Participants responses are measured using the mean score on the 9-item visual analogue scales, with 100-mm lines, with 0 representing the best outcome and 100 representing the worst outcome.
Time Frame: Up to 6 months
Population: Quality of Life parameters were to be analyzed in Part 2 of the study. Due to low enrollment, the study was terminated early and Part 2 was not performed.
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to 28 Days (AUC0-28d) of Sotatercept Following a Single Dose
Description: AUC0-28d is a measure of the mean concentration levels of a drug in the plasma from time 0 to 28 days.
Time Frame: Pre-dose 1 Day 1, 4 hours post-dose Day 1, Day 5, Day 8, Day 11, Day 15, Day 22, Day 28
Population: All participants who received at least 1 dose of study treatment and had data for AUC0-28d of Sotatercept Following a Single Dose
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 13 | 7
day*ng/mL | 24443.28 (8130.52) | 43977.03 (18490.17)

9. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Infinity (AUC0-inf) of Sotatercept Following a Single Dose
Description: AUC0-inf is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time.
Time Frame: Pre-dose 1 Day 1, 4 hours post-dose Day 1, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 36, pre-dose 2 Day 43
Population: All participants who received at least 1 dose of study treatment and had data for AUC0-inf of Sotatercept Following a Single Dose
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 10 | 3
day*ng/mL | 40145.34 (20680.76) | 137994.6 (18183.66)

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Sotatercept Following a Single Dose
Description: Cmax is a measure of the maximum amount of drug in the plasma after a dose is given.
Time Frame: Pre-dose 1 Day 1, 4 hours post-dose Day 1, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 36, pre-dose 2 Day 43
Population: All participants who received at least 1 dose of study treatment and had data for Cmax of Sotatercept Following a Single Dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 14 | 9
ng/mL | 1325.33 (435.89) | 2069.68 (842.43)

11. Secondary Outcome: Time to Maximum Concetration (Tmax) of Sotatercept Following a Single Dose
Description: Tmax is a measure of the time it takes for a drug to reach maximum concentration in the plasma after the dose is given.
Time Frame: Pre-dose 1 Day 1, 4 hours post-dose Day 1, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 36, pre-dose 2 Day 43
Population: All participants who received at least 1 dose of study treatment and had data for Tmax of Sotatercept Following a Single Dose of Sotatercept
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 14 | 9
Days | 8.16 (3.78) | 12.31 (7.67)

12. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Sotatercept Following a Single Dose
Description: t1/2 is the elimination half-life of study drug: the time it takes for half of the study drug in the blood plasma to dissipate.
Time Frame: Pre-dose 1 Day 1, 4 hours post-dose Day 1, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 36, pre-dose 2 Day 43
Population: All participants who received at least 1 dose of study treatment and had data for t1/2 of Sotatercept Following a Single Dose
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 10 | 3
Days | 18.98 (7.96) | 30.84 (9.46)

13. Secondary Outcome: Apparent Serum Clearance (CL/F) of Sotatercept Following a Single Dose
Description: Apparent serum CL is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose 1 Day 1, 4 hours post-dose Day 1, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 36, pre-dose 2 Day 43
Population: All participants who received at least 1 dose of study treatment and had data for CL/F of Sotatercept Following a Single Dose
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 10 | 3
mL/day | 479.36 (254.44) | 220.14 (31.17)

14. Secondary Outcome: Apparent Volume of Distribution (Vz/F) Following a Single Dose of Sotatercept
Description: Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: Pre-dose 1 Day 1, 4 hours post-dose Day 1, Day 5, Day 8, Day 11, Day 15, Day 22, Day 29, Day 36, pre-dose 2 Day 43
Population: All participants who received at least 1 dose of study treatment and had data for Vz/F of Sotatercept Following a Single Dose
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
Number analyzed (Participants) | 10 | 3
mL | 11944.60 (7172.84) | 9849.80 (3449.33)

ADVERSE EVENTS:
Time Frame: Up to approximately 6 months
Description: The safety analysis population included all participants who received at least one dose of study treatment. The analysis population for All-Cause Mortality included all enrolled participants.
Arm/Group | Sotatercept 15 mg | Sotatercept 30 mg
All-Cause Mortality (participants affected / at risk) | 6/14 | 5/12
Serious Adverse Events (participants affected / at risk) | 4/14 | 8/11
Other Adverse Events (participants affected / at risk) | 14/14 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept 15 mg (N=14) | Sotatercept 30 mg (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept 15 mg (N=14) | Sotatercept 30 mg (N=11)
Anaemia (Blood and lymphatic system disorders) | 4 (34) | 6 (17)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (23) | 4 (9)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (28) | 5 (21)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Ocular icterus (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Caecitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9) | 1 (1)
Poor dental condition (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 2 (4) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (14) | 4 (6)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 4 (9) | 4 (6)
Pyrexia (General disorders) | 1 (1) | 1 (2)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (4)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Lymph node palpable (Investigations) | 1 (2) | 0 (0)
Protein total decreased (Investigations) | 1 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (2)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (22) | 4 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (9) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (24) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (5) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (19) | 3 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4) | 2 (6)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2)
Feeling of despair (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tobacco user (Social circumstances) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 2 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT01284348/Prot_SAP_000.pdf